CLINICAL TRIAL: NCT00364507
Title: Serum Levels of Insulin-Like Growth Factor in Fertile and Infertile Women Over 40 Years Old
Brief Title: Serum Levels of Insulin- Like Growth Factor and Fertility
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: IGF1-HMO-CTIL
Record Dates: First submitted 2006-08-14; First posted 2006-08-15 (Estimated); Last update posted 2006-08-15 (Estimated); Status verified 2006-08

CONDITIONS: Fertility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
this study will try to determine whether serum levels of insulin like growth factor are higher in fertile women than infertile women.

DETAILED DESCRIPTION:
this study will try to determine whether serum levels of insulin like growth factor are higher in fertile women than infertile women.The women will over 40 years old.

ELIGIBILITY:
Inclusion Criteria:

* 40-55 years old
* healthy

Exclusion Criteria:

* pregnant women
* breast feeding
* menopause
* vegetarian

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-01; Study Completion 2007-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: David MANKUTA, MD, Study Chair — Hadassah Medical Orginization